CLINICAL TRIAL: NCT00340717
Title: Multi-Institutional Pilot Study to Evaluate Molecular Markers in Urine and Serum in the Early Detection of Prostate Cancer
Brief Title: Markers for Early Detection of Prostate Cancer
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999903187; 03-C-N187
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-09

CONDITIONS: Prostate Cancer
Keywords: Methylation; Genes; Screening; Prospective; Diagnosis
MeSH Terms: conditions — Prostatic Neoplasms; Disease

SUMMARY:
This study will determine whether certain gene alterations can serve as markers for early detection of prostate cancer. Prostate cancer is often diagnosed by detecting high levels of a protein called prostate-specific antigen (PSA) in the blood. Other conditions can also cause elevated PSA levels, however, so that additional tests are needed to distinguish between benign and cancerous prostate conditions.

Patients between 40 and 75 years of age who are referred to Howard University Hospital in Washington, D.C., or Madigan Army Medical Center in Tacoma, Washington, for ultrasound and needle biopsy to diagnose prostate cancer may be eligible for this study.

Participants will undergo the following procedures at the time of the biopsy visit:

* Blood collection: Patients have 10 milliliters (2 teaspoons) of blood drawn.
* Prostate massage: Patients have a rectal examination and prostate massage. For the latter procedure, the physician lightly massages the prostate gland for about 15 seconds. After the massage, the patient provides a urine specimen.
* Biopsy: A small sample of tumor tissue is removed surgically for examination under the microscope.

Patients whose initial biopsy does not show cancer cells, but who are advised to have a repeat biopsy in the future will give a blood, urine, and biopsy specimen at the time of the next biopsy.

Patients who are diagnosed with prostate cancer and undergo surgery to remove the tumor will have a small sample of tumor tissue set aside for this study to look for substances that may help predict prostate cancer.

DETAILED DESCRIPTION:
In the U.S., screening by prostate-specific antigen (PSA) is widespread and considered to be an effective early detection screen for prostate cancer although there are some problems associated with its use. Only about 30-40% of men with elevated PSA are diagnosed with cancer on initial biopsy. The other 60-70% are diagnosed with either benign prostatic hyperplasia or low-or high-grade prostatic intraepithelial neoplasia (LGPIN or HGPIN). Due to their persistent elevated PSA levels, men undergo repeat biopsies where many are subsequently diagnosed with cancer (the false negative rate for biopsies with pathological diagnoses of benign or LGPIN has been reported to be 13-19% and for HGPIN from 50-70%). We propose to conduct a pilot study to evaluate whether (i) the addition of molecular markers (e.g., tumor-specific gene methylation of GSTPI, CD44, Annexin II, and Caveolin 1) detectable in serum and/or urine sediments after prostatic massage can improve the prediction of prostate cancer and (ii) addition of tumor-specific gene methylation detectable in core-needle biopsy specimens can improve the sensitivity of core-needle biopsy in the diagnosis of prostate cancer among patients screened at two Urology clinics located at Howard University, Washington, DC and Madigan Army Medical Center, Tacoma, WA. Preliminary studies have shown detection of hypermethylated genes in urine sediments after prostatic massage in men with elevated PSA (greater than 4ng/ml) improved the specificity of PSA from 73% to 98%. Further, DNA hypermethylation of tumor-specific genes was also identified in serum. In our laboratory, we have developed assays for evaluating DNA hypermethylation of several genes shown to be important in prostate carcinogenesis. These assays are highly sensitive (able to detect down to about 20 tumor cells with methylated DNA) and specific (can distinguish methylated from normal DNA from in a ratio of 1 tumor cell in 10,000 normal cells), and could serve to add value to current prostate cancer screening modalities.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must be within 40-75 years of age.

Patients referred for diagnostic transrectal ultrasound and prostate needle biopsy.

Patients must be adults and capable of understanding and signing an informed consent form.

Patients must be willing to undergo a brief prostatic massage and provide a urine and serum specimen prior to diagnostic core needle biopsy.

EXCLUSION CRITERIA:

Patients with active of history of other malignancy (excluding non-melanoma skin cancer).

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2003-05

CONTACTS AND LOCATIONS:
Locations (1):
- Madigan Army Medical Center, Tacoma, Washington, United States

REFERENCES:
- [Background] Orozco R, O'Dowd G, Kunnel B, Miller MC, Veltri RW. Observations on pathology trends in 62,537 prostate biopsies obtained from urology private practices in the United States. Urology. 1998 Feb;51(2):186-95. doi: 10.1016/s0090-4295(97)00620-1. PMID 9495696